CLINICAL TRIAL: NCT03972059
Title: The Effect of High Intensity Interval Circuit Training With Portable Equipment on Changes in Resting Metabolic Rate in Overweight Adults
Brief Title: High Intensity Interval Circuit Training on Resting Metabolic Rate in Overweight Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HIICT-RMR study
Record Dates: First submitted 2019-05-23; First posted 2019-06-03 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Intervention Model Description: The 12-week training program will be divided into 3 phases (4 weeks each phase). Completion of each phase means that the subjects have increased their physical fitness and will get to the next phase where the intensity of exercise will increase in order to gain more physical fitness benefits (e.g. increased caloric expenditure). There will be a control group as well, where participants will not participate in any intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): A 12-week high intensity interval circuit training program for weight management in overweight adults.
  Interventions: Other: Exercise training - Phase 1; Other: Exercise training - Phase 2; Other: Exercise training - Phase 3
- Control group (No Intervention): No intervention for 12 weeks, participants perform all tests.

INTERVENTIONS:
Other: Exercise training - Phase 1 — Phase 1 is the first 4 weeks of the 12-week training program.
  Arms: Experimental group
Other: Exercise training - Phase 2 — Phase 2 is the next 4 weeks following phase 1 of the 12-week training program. The exercise intensity during exercise bouts in this phase is increased compared to the exercise intensity applied in phase 1.
  Arms: Experimental group
Other: Exercise training - Phase 3 — Phase 3 is the last 4 weeks of the 12-week training program. The exercise intensity during exercise bouts in this phase is increased compared to the exercise intensity applied in the previous phases.
  Arms: Experimental group

SUMMARY:
This is the first study to examine changes in resting metabolic rate up to 72 hours following an exercise session, and how these changes may be affected by 12 weeks of high intensity interval circuit training (HIICT). Various training programs that have been implemented in previous studies have investigated changes in resting metabolic rate only for the first 2-8 hours following an exercise session.

Briefly, the results of this study will provide insight into the following:

1. To what extent and for how long does HIICT increases the resting metabolic rate following an exercise session?
2. How can this exercise program enhance metabolism without any dietary or other exercise intervention?
3. What is the caloric deficit that will result from 3 months of HIICT and how to what extent this deficit will influence body weight reduction?

DETAILED DESCRIPTION:
According to the World Health Organization, overweight and obesity are defined as as abnormal or excessive fat accumulation, that presents a risk to health. Body Mass Index (BMI) is a useful population-level measure of overweight and obesity in adults, defined as follows: BMI = [weight (kg)] / [height (m)^2]. Individuals with BMI>25 kg/m^2 are considered overweight, whereas individuals with BMI>30 are considered obese. The higher the BMI, the greater the risk of developing non-communicable diseases, such as cardiovascular disease, diabetes mellitus and various forms of cancer. Obesity is now the most widespread disease in the developed world. It has been estimated that over 1.9 billion adults (39% of the population) are overweight, of whom 600 million (13% of the population) are obese. These rates are translated into a significant economic impact on a county's health care system; therefore, drastic measures are needed. The major cause of obesity is an energy imbalance between caloric intake and energy expenditure in favor of the former. Thus, changes in lifestyle that affect the energy balance, such as participation in an exercise program, can reduce body weight and, therefore, contribute to obesity treatment.

The recommendation of physical activity for significant weight loss involves prolonged exercise of moderate to high intensity that gradually increases to ~250 minutes/week. Resistance training is also recommended as it activates the neuromuscular system and can improve functional ability. On the other hand, High Intensity Interval Training (HIIT), which mainly involves a cardiovascular exercise strategy alternating short periods of intense anaerobic exercise with less intense recovery periods, are proposed because they are time-efficient. In addition, HIIT improves aerobic capacity and body composition, which is related to resting metabolic rate and mitochondrial metabolism of skeletal muscle in both healthy and overweight and obese adults. Changes caused by HIIT in mitochondrial function may explain the greater efficacy in inducing positive metabolic adaptations compared to traditional endurance or resistance protocols, even when not accompanied by dietary weight loss strategies.

Resting metabolic rate is defined as the energy expenditure required to maintain the normal physiological processes of the body at rest and accounts for 60-75% of the total daily energy expenditure. Small increases in resting metabolic rate could long-term positive effects on weight management. Energy expenditure is increased not only during exercise, but also for some hours post-exercise. To date, it has been observed that this increase in resting metabolic rate can last for up to 48 hours following an exercise session, especially following resistance training. More specifically, in a study where 7 women (22-35 years old) participated in a resistance training program (100 minutes/session, 10 exercises of 5 sets with 10-15 repetitions per set), there was an increase in their resting metabolic rate by 13% at the first 3 hours and an increase by 4.2% at 16 hours following an exercise session. On the other hand, a 10-week (3 session/week) strength training program with an intensity of 65-85% of the maximum heart rate based on age (gradual increase in intensity), did not appear to cause any changes in resting metabolic rate following an exercise session. However, in another study where resistance training (strength protocol of 3 sets with 10-15 repetitions per set at the beginning of intervention up to 4-8 repetitions at the end of the intervention) was combined with endurance training (65% to 85% with an intensity of 65-85% of the maximum heart rate based on age, of increasing intensity), it was observed that resting metabolic rate increased following an exercise session.

It is important to note that, according to the available literature, it has been shown that training studies have been examined changes in resting metabolic rate only up to 2-8 hours following an exercise session. Therefore, the aim of the present study is to investigate the effect of a 12-week HIICT protocol with portable equipment on changes in resting metabolic rate 24, 48 and 72 hours following an exercise session.

Flow of the research design:

1. Baseline: Anthropometric and physiological measurements (including a Resting Metabolic Rate (RMR) measurement following an overnight fast).
2. One-week familiarization period: Volunteers will participate in two exercise sessions in order to learn the right techniques. RMR will be measured 24, 48 and 72 hours following the last exercise session. Moreover, participants will be given instructions and then they will record their diet for 3 days (2 week days and one weekend day).
3. Initiation of the 12-week HIICT program: The program will be supervised and portable training equipment will be used. There will be 3 exercise sessions per week (Monday-Wednesday-Friday). The program will be divided into 3 phases (4 weeks each phase), where exercise intensity will increase gradually.
4. 1st phase: RMR will be measured 24 hours before, as well as 24, 48 and 72 hours following the last exercise session of the phase (e.g. at the end of the 4th week of the program). Anthropometric and physiological measurements will also be conducted. Moreover, participants will record their diet for 3 days (2 week days and one weekend day).
5. 2nd phase: Exercise intensity will increase. The same measurements with phase 1 will be conducted.
6. 3rd phase: Exercise intensity will increase. The same measurements with phases 1 and 2 will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or class I obesity (BMI: 25-35 kg/m^2)
* Sedentary lifestyle
* Willing to lose weight
* Individuals at low risk of various cardiovascular, pulmonary, renal, and metabolic diseases as well as other conditions (e.g., pregnancy and orthopedic injury) that require special attention when developing the exercise prescription (Thompson et al., 2013). This risk classification indicates that participants will be able to participate in moderate intensity exercise [40-60% oxygen uptake reserve (VO2R); 3-6 metabolic equivalent of task (METs)] and also in vigorous intensity exercise (>60% VO2R; >6 METs) while medical examination, exercise test and physician supervision are not recommended in the preparticipation health screening process.

Exclusion Criteria:

* Following a diet plan or taking dietary supplements over the last 6 months and during the intervention
* Participation in another training program over the last 6 months and during the intervention
* Family history of coronary heart disease
* Recent musculoskeletal injury

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Resting metabolic rate (kilocalories) | At baseline
  Resting metabolic rate following 12 hours of an overnight fast
Resting metabolic rate (24 before an exercise bout) (kilocalories) | Pre-intervention, 24 hours after completion of phase 1, 24 hours after completion of phase 2, 24 hours after completion of phase 3
  Changes in resting metabolic rate 24 before an exercise bout
Resting metabolic rate (24 following an exercise bout) (kilocalories) | Pre-intervention, 24 hours after completion of phase 1, 24 hours after completion of phase 2, 24 hours after completion of phase 3
  Changes in resting metabolic rate 24 following an exercise bout
Resting metabolic rate (48 following an exercise bout) (kilocalories) | Pre-intervention, 24 hours after completion of phase 1, 24 hours after completion of phase 2, 24 hours after completion of phase 3
  Changes in resting metabolic rate 48 following an exercise bout
Resting metabolic rate (72 following an exercise bout) (kilocalories) | Pre-intervention, 24 hours after completion of phase 1, 24 hours after completion of phase 2, 24 hours after completion of phase 3
  Changes in resting metabolic rate 72 following an exercise bout
Body fat mass (kilograms) | At baseline, 24 hours after completion of phase 1, 24 hours after completion of phase 2, 24 hours after completion of phase 3
  Changes in body fat mass measured with dual-energy x-ray absorptiometry (DEXA)
Body lean mass (kilograms) | At baseline, 24 hours after completion of phase 1, 24 hours after completion of phase 2, 24 hours after completion of phase 3
  Changes in body lean mass measured with dual-energy x-ray absorptiometry (DEXA)
Bone mass (kilograms) | At baseline, 24 hours after completion of phase 1, 24 hours after completion of phase 2, 24 hours after completion of phase 3
  Changes in bone mass measured with dual-energy x-ray absorptiometry (DEXA)

SECONDARY OUTCOMES:
Waist to hip ratio (WHR) | At baseline, 24 hours after completion of phase 1, 24 hours after completion of phase 2, 24 hours after completion of phase 3
  WHR is calculated by dividing waist circumference by hip circumference
Lower limb strength | At baseline, 24 hours after completion of phase 1, 24 hours after completion of phase 2, 24 hours after completion of phase 3
  Leg press (10 Repetition Maximum - RM)
Upper body strength | At baseline, 24 hours after completion of phase 1, 24 hours after completion of phase 2, 24 hours after completion of phase 3
  Chest press (10 Repetition Maximum - RM)
Aerobic capacity test | At baseline, 24 hours after completion of phase 1, 24 hours after completion of phase 2, 24 hours after completion of phase 3
  Ebbeling submaximal treadmill walking test
Maximal abdominal muscle endurance | At baseline, 24 hours after completion of phase 1, 24 hours after completion of phase 2, 24 hours after completion of phase 3
  Maximal repetition till exhaustion

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis G Fatouros, PhD, Study Director — SmArT Lab, DPESS, University of Thessaly
Locations (1):
- SmArT LABORATORY, SCHOOL OF PHYSICAL EDUCATION & SPORTS SCIENCES, UNIVERSITY OF THESSALY, Trikala, Greece

IPD SHARING:
Plan to Share IPD: No